CLINICAL TRIAL: NCT06972615
Title: A Phase II, Single Arm Study, Evaluating Intravesical Gemcitabine/Docetaxel in Combination With Systemic Pembrolizumab in Subjects With High Risk NMIBC Unresponsive to BCG Therapy
Brief Title: Intravesical Chemotherapy in Combination With Systemic Pembrolizumab in NMIBC Unresponsive to BCG Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BLATAM (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-G14
Record Dates: First submitted 2025-04-18; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): intrravesical docetaxel plus gemcitabine and intravenous pembrolizumab
  Interventions: Drug: intravesical Chemotherapy docetaxel/gemcitabine

INTERVENTIONS:
Drug: intravesical Chemotherapy docetaxel/gemcitabine — intravesical quimiotherapy plus intravenous immunotherapy
  Other Names: pembrolizumb

SUMMARY:
interventional study of intravesical chemotherapy and sistemic immunotherapy in NMIBC

DETAILED DESCRIPTION:
patients will receive intrravesical chemotherapy every 3 weeks and systemic pembrolizumb every 6 week. for a total of 1 year of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide documented informed consent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
2. Be ≥18 years of age on the day of signing informed consent.
3. Have a histologically confirmed diagnosis of high-risk non-muscle invasive (T1, High Grade Ta and/or CIS) transitional cell carcinoma of the bladder. Subjects with tumors of mixed transitional/non-transitional cell histology are allowed, but transitional cell carcinoma must be the predominant histology. Subjects with predominant or exclusively non-transitional cell histology are not allowed. Confirmation of histology, grade and stage will be performed by central review and must be completed during the screening period and prior to enrollment.
4. In subjects who have papillary tumors (Ta and T1), a complete TURBT must have been performed, as characterized by:Attainment of a visually complete resection of all papillary tumors (Ta and T1) 5- Have been treated with adequate BCG therapy and have developed high risk NMIBC that is unresponsive or exposed to BCG therapy.

Adequate BCG therapy must include:

* An induction course with at least 5 out of 6 BCG instillations (adequate induction); and
* At least 7 out of 9 BCG instillations within 9 months of the first instillation of adequate induction therapy

BCG unresponsive high risk NMIBC is defined as:

* Stage progression at 3 months (±4 weeks) despite adequate induction therapy (e.g., Ta to T1, or CIS to T1; note: adequate induction therapy only, defined above, is required in this case); or
* High grade T1 disease at the first evaluation after adequate BCG induction or
* Persistent high risk NMIBC at 6 months (±4 weeks) after adequate BCG; or
* Recurrent high risk NMIBC within 12 months of the last BCG instillation despite having received adequate BCG.

BCG Exposed is defined as: having high-grade persistent (BCG resistant) or recurrent NMIBC within 24 months of the last BCG dose but not meeting the definition of BCG-unresponsive

Exclusion Criteria:

* 1. Has muscle-invasive (i.e. T2, T3, T4) locally advanced non-resectable or metastatic urothelial carcinoma.

  2. Has concurrent extra-vesical (i.e. urethra, ureter or renal pelvis) non-muscle-invasive transitional cell carcinoma of the urothelium.

  3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

  4. Has undergone any intervening intravesical chemotherapy or immunotherapy from the time of most recent cystoscopy/ transurethral resection of bladder tumor to starting trial treatment. (Note: A single dose of intravesical treatment given as part of the most recent cystoscopy/ transurethral resection of bladder tumor, during the screening period, such as with chemotherapy as per local/regional practices, is acceptable.)

  5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1, Day 1 or who has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
eficacy | 3 months
  Complete Response rate
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  To evaluate safety and tolerability of systemic pembrolizumab in combination with intravesical gemcitabine/docetaxel

CONTACTS AND LOCATIONS:
Locations (1):
- BLATAM, CABA, Argentina

IPD SHARING:
Plan to Share IPD: Yes
de-identified demographic information (age, sex), baseline disease characteristics, treatment received, key efficacy outcomes (e.g., response rates, progression-free survival, overall survival), and safety data (adverse events). Data will be shared in aggregate or de-identified format to ensure patient confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1/jun/2025
Access Criteria: data will be available on web site

REFERENCES:
- See also: Related Info — https://blatam.com/